CLINICAL TRIAL: NCT00708643
Title: Clinical Performance of a New Daily Disposable Contact Lens Worn in an Established Contact Lens Wearing Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-0803
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2010-12-01 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Refractive Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Habitual silicone hydrogel (Active Comparator): Habitual contact lens wear.
  Interventions: Device: Habitual Silicone Hydrogel Contact Lens
- narafilcon A (Experimental): Silicone hydrogel daily disposable contact lens
  Interventions: Device: narafilcon A

INTERVENTIONS:
Device: Habitual Silicone Hydrogel Contact Lens — contact lens
  Arms: Habitual silicone hydrogel
Device: narafilcon A — contact lens
  Arms: narafilcon A

SUMMARY:
This study seeks to evaluate the clinical and subjective performance of a new daily disposable soft contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (17 years) and capacity to volunteer.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
5. They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
6. They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
7. They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
10. They have diabetes.
11. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Started | 40 | 40
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Includes all subjects that completed the study.
  years | 28.3 (9.9) | 25.8 (8.7) | 27.2 (9.6)
Gender [Number; unit: participants] — Includes all subjects that completed the study.
  participants
    Female | 32 | 33 | 65
    Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants] — Includes all subjects that completed the study.
  participants
    Canada | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Limbal Hyperemia
Description: Measures the redness of the limbal region of the eye on a scale of 0 to 100 grade with 0=none and 100=severe. The analysis is the average grade over all time frames.
Time Frame: At 2 weeks and 4 weeks
Population: The analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale | 34.0967 (1.4982) | 31.0920 (1.7271)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; The alternative hypothesis is that narafilcon A will provide a lower level of limbal hyperemia than the habitual lens; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -3.0047, 98.75% CI 2-sided [-3.0047 to 2.7153], Standard Error of Mean 2.2863 — The mean difference is calculated as narafilcon A minus the habitual lens

2. Primary Outcome: Lens Comfort
Description: Rating of lens comfort by rating agreement to the following statement:
  "The lenses I am wearing are comfortable."
  Rating using the following scale:
  1=strongly agree, 2=agree, 3=neutral, 4=disagree, 5=strongly disagree. The rating is averaged over all time frames.
Time Frame: At 3,7,10,13,17,21,24, and 27 days
Population: The analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale | 1.1078 (0.4993) | 1.0274 (0.5737)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; The alternative hypothesis is that narafilcon A provides better comfort than the habitual lens by having a lower rating on the scale; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.0804, 99% CI 2-sided [-0.0804 to 1.8821], Standard Error of Mean 0.7605 — The mean difference is calculated as narafilcon A minus habitual lens

3. Primary Outcome: Upper Lid Margin Staining
Description: Measures the trauma to tissue that lines the margin of the inside of the upper eyelid on a 0 to 3 scale, with 0=none to 3=severe. The analysis is the average grade over all time frames.
Time Frame: At 2 weeks and 4 weeks.
Population: The analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale.
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale. | 0.9358 (1.1146) | 1.1586 (1.2857)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; The alternative hypothesis is that narafilcon A provides a lowe level of upper lid margin staining than the habitual lens; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.2228, 99% CI 2-sided [0.2228 to 4.6564], Standard Error of Mean 1.7002 — The mean difference is calculated as narafilcon A minus the habitual lens

4. Secondary Outcome: Tarsal Roughness
Description: Measures the amount of roughness to the tissue of the inside upper and lower eyelid on a scale of 0 to 100 with 0=none and 100=severe. The analysis is the average grade over all time frames.
Time Frame: At 2 weeks and 4 weeks
Population: The analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale | 30.1028 (0.7784) | 31.3624 (0.8994)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.2596, 98.75% CI 2-sided [1.2596 to 4.2599], Standard Error of Mean 1.1873 — The mean difference is calculated as narafilcon A minus the habitual lens

5. Secondary Outcome: Tarsal Hyperemia
Description: Measures the amount of redness to the tissue of the inside upper and lower eyelid using a 0 to 100 scale with 0=none and 100=severe.
Time Frame: At 2 weeks and 4 weeks.
Population: The analysis includes all subjects that completed the study.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale | 38.4103 (1.5238) | 37.5478 (1.7646)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; The alternative hypothesis is that narafilcon A provides a lower level of tarsal hyperemia than the habitual lens; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.8625, 98.75% CI 2-sided [-0.8625 to 5.0524], Standard Error of Mean 2.3407 — The mean difference is calculated as narafilcon A minus habitual lens

6. Secondary Outcome: Corneal Staining
Description: A measure of corneal abrasion using a 0 to 100 scale with 0=none, 25=micropunctate, 50=macropunctate, 75=coalescence, 100=patch. The analysis is the average grade over all time frames.
Time Frame: At 2 weeks and 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Number analyzed (Participants) | 40 | 39
units on a scale | 6.6173 (1.1106) | 6.3763 (1.2820)
Statistical Analysis 1: Comparison: Habitual Silicone Hydrogel vs Narafilcon A; The alternative hypothesis is that narafilcon A provides lower levels of corneal staining than the habitual lens; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.2410, 98.75% CI 2-sided [-0.2410 to 4.0043], Standard Error of Mean 1.6975 — The mean difference is calculated as narafilcon A minus habitual lens

ADVERSE EVENTS:
Arm/Group | Habitual Silicone Hydrogel | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.